CLINICAL TRIAL: NCT07196878
Title: Ultrasound-Guided Percutaneous Neuromodulation Protocol to Improve Gait Rehabilitation in Patients Who Have Suffered a Stroke. Clinical Trial.
Brief Title: Percutaneous Ultrasound-guided Neuromodulation to Improve Gait Rehabilitation in Patients Who Have Suffered a Stroke.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alejandro Martín García (Other)
Responsible Party: Sponsor-Investigator, Alejandro Martín García, Ultrasound-Guided Percutaneous Neuromodulation Protocol to Improve Gait Rehabilitation in Patients Who Have Suffered a Stroke. Clinical Trial., Universidad de Zaragoza
Organization: Universidad de Zaragoza (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C.I. PI25/059
Record Dates: First submitted 2025-09-19; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Ictus; Gait Disorders, Neurologic
Keywords: ICTUS; Gait disorder; Ultrasound guided neuromodulation
MeSH Terms: conditions — Gait Disorders, Neurologic; Mobility Limitation

STUDY DESIGN:
Intervention Model Description: An intervention group receiving the procedure in addition to their usual treatment is compared with a control group that receives only their usual treatment (the same as the intervention group).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound-Guided Percutaneous Neuromodulation (Experimental): Ultrasound-guided percutaneous neuromodulation is performed 10 times, each lasting 10 seconds with 10-second rest intervals.
  Interventions: Other: Ultrasound-Guided Percutaneous Neuromodulation
- Control group (No Intervention): Control group that does not receive the intervention; it is used solely for comparison.

INTERVENTIONS:
Other: Ultrasound-Guided Percutaneous Neuromodulation — An ultrasound-guided puncture is performed to place one needle near the sciatic nerve and another near the peroneal nerve. Then, an electrical stimulus at 10 Hz is applied for 10 seconds, repeated 10 times.
  Arms: Ultrasound-Guided Percutaneous Neuromodulation

SUMMARY:
The goal of this clinical trial is to learn if percutaneous ultrasound-guided neuromodulation (NMP-e) can improve gait rehabilitation in adults who have suffered a stroke. The main questions it aims to answer are:

* Does NMP-e improve walking speed in stroke survivors?
* Does NMP-e enhance muscle strength, functional mobility, reduce spasticity, improve balance, and increase health-related quality of life?

Researchers will compare the addition of NMP-e to conventional physiotherapy versus conventional physiotherapy alone to see if the intervention provides additional benefits in gait rehabilitation and other functional outcomes.

Participants will:

* Continue their regular physiotherapy treatment consisting of passive and active-assisted mobilizations and strength exercises.
* Receive NMP-e targeting the sciatic nerve at mid-thigh and the common peroneal nerve at the fibular head (experimental group only).
* Undergo stimulation with an electrostimulator at 10 Hz for 10 seconds per trial, repeated 10 times, with intensity adjusted for comfort.
* Be evaluated before the intervention, immediately after, and one week later using:
* 10-Meter Walk Test for gait speed
* Dynamometry for ankle plantarflexor and dorsiflexor strength
* Time Up and Go test for functional mobility
* Modified Modified Ashworth Scale for spasticity
* Berg Balance Scale for balance
* EuroQoL-5 Dimensions for health-related quality of life

Participants must be adults aged 18-70, able to walk 10 meters without assistance, currently receiving physiotherapy, and able to provide informed consent. Key exclusions include pregnancy, bleeding disorders, needle allergies, systemic inflammatory disorders, or recent invasive physiotherapy.

This randomized controlled trial will be conducted at ATECE, **a Spanish association dedicated to the care and rehabilitation of individuals with acquired brain injury**, where participants will be recruited and receive their interventions. The study aims to evaluate the potential of NMP-e as an adjunctive therapy for improving gait and related functional outcomes in subacute and chronic stroke patients.

DETAILED DESCRIPTION:
This study is designed to evaluate the effectiveness of ultrasound-guided percutaneous neuromodulation (PNM) combined with conventional physiotherapy in improving gait and functional outcomes in adults recovering from subacute to chronic stroke. Stroke is a leading cause of long-term disability worldwide, frequently resulting in impaired motor control, reduced muscle strength, altered gait patterns, and decreased functional independence. Conventional physiotherapy remains the cornerstone of post-stroke rehabilitation, focusing on exercises to enhance strength, coordination, balance, and mobility. However, recovery is often incomplete, and additional interventions that can augment neuroplasticity and motor recovery are critically needed.

Ultrasound-guided PNM is a minimally invasive technique that involves targeted electrical stimulation of peripheral nerves via a fine needle under ultrasound guidance. By stimulating the sciatic and deep peroneal nerves, PNM may enhance neuromuscular activation, improve muscle recruitment, reduce spasticity, and facilitate motor relearning. This trial seeks to determine whether integrating PNM with standard physiotherapy produces greater improvements in walking speed, lower limb strength, balance, and functional mobility compared to physiotherapy alone.

A total of 30 participants aged 18-70 years who have experienced a stroke at least three months prior and are capable of walking a minimum of 50 meters with or without assistive devices will be enrolled. Participants will be randomly assigned in a 1:1 ratio to either the experimental group, receiving ultrasound-guided PNM plus physiotherapy, or the control group, receiving physiotherapy alone. The intervention will be delivered over multiple sessions following a standardized protocol. In the experimental group, the PNM sessions will target the sciatic and deep peroneal nerves of the affected limb, using a pre-determined stimulation frequency and intensity individualized to each participant's tolerance. Physiotherapy sessions will include strength training, gait training, balance exercises, and functional mobility tasks, applied consistently across both groups.

Outcomes will be assessed at baseline, immediately post-intervention, and one week after the last treatment session to capture both immediate and short-term effects. The primary outcome measure is walking speed, assessed using the 10-Meter Walk Test, a validated and widely used metric of functional gait performance. Secondary outcomes include lower limb muscle strength (ankle dorsiflexors and plantarflexors) measured with handheld dynamometry, spasticity assessed by the Modified Modified Ashworth Scale, functional mobility evaluated using the Timed Up and Go test, balance assessed with the Berg Balance Scale, and health-related quality of life measured with the EQ-5D questionnaire.

Data will be analyzed using mixed linear and logistic regression models, accounting for repeated measures and individual variability. Safety and tolerability will be closely monitored throughout the study, with adverse events recorded and managed according to established protocols. Participants will provide informed consent and retain the right to withdraw from the study at any time without any consequences to their ongoing care.

This trial aims to provide robust evidence regarding the potential additive benefits of ultrasound-guided PNM to conventional physiotherapy in post-stroke rehabilitation. Demonstrating a significant improvement in gait, muscle strength, and functional independence could support the adoption of PNM as a novel, evidence-based adjunct therapy for stroke survivors, potentially enhancing long-term outcomes and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Be between 18 and 70 years of age;
2. Have suffered a stroke (CVA);
3. Be in the subacute or chronic phase of the disease;
4. Be able to walk 10 meters without assistance from another person;
5. Currently be undergoing physiotherapy with conservative techniques;
6. Be able to understand the technique being applied;
7. Sign the informed consent form.

Exclusion Criteria:

1. Belonephobia (fear of needles);
2. Allergy to needles or metals;
3. Presence of uncontrolled coagulopathies;
4. Presence of uncontrolled arterial disease;
5. Pregnancy;
6. Dermatological disorders;
7. Presence of diseases such as systemic inflammatory disorders (e.g., rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, or septic arthritis);
8. Presence of diseases such as tumors, cancer, or metastases;
9. Having received invasive physiotherapy treatment in the last 4 weeks.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Velocidad | This variable will be measured before, immediately after, and one week later.
  The speed will be measured using the 10-Meter Walk Test.

SECONDARY OUTCOMES:
Isometric strength of the ankle plantarflexor and dorsiflexor muscles. | It will be measured before, immediately after, and one week following the intervention.
  The strength of the ankle flexor and extensor muscles will be measured using a dynamometer.
Functional mobility will be assessed using the Timed Up and Go (TUG) test. | The measurement will be taken before, immediately after, and one week following the intervention.
  The participant will be seated in a chair until they hear the evaluator's signal to start the test. The participant must stand up, walk a total of 3 meters in a straight line, return to the chair, and resume the starting position. Three measurements will be taken, and the best result will be considered the most accurate.
Spasticity will be assessed using the Modified Modified Ashworth Scale (MMAS). | It will be measured before, immediately after, and one week following the intervention.
  Muscle tone of the hamstring and anterior tibial muscles will be measured.
Balance will be assessed using the Berg Balance Scale (BBS). | It will be measured before, immediately after, and one week following the intervention.
  Participants will perform a total of 14 tasks, which include: standing up from a seated position, maintaining a standing position without support, sitting without leaning the back while keeping the feet on the floor or on a footrest, sitting down from a seated position, performing two transfers from one chair to another and returning to the first chair, maintaining a standing position without support with eyes closed, maintaining a standing position without support with feet together, reaching forward with an extended arm, picking up an object from the floor while standing, turning the head backward over the right and left shoulders while standing, performing a 360º turn, alternately stepping one foot onto a step or footrest while standing without support, maintaining a standing position without support with one foot forward, and maintaining a one-legged stance.
Health-related quality of life will be assessed using the EuroQoL-5 Dimensions (EQ-5D) scale. | The scale will be administered before, immediately after, and one week following the intervention.
  It consists of two main parts: the first is a description of the individual's health across five domains, and the second is the Visual Analog Scale (VAS), which assesses the individual's overall perception of health. The first part of the scale evaluates: a) mobility; b) self-care; c) usual activities; d) pain/discomfort; e) anxiety/depression. Each domain has five response levels describing the degree of difficulty experienced by the individual, ranging from no difficulty to extreme difficulty. The second part is assessed using a line on which the individual marks their overall perception of health at the time of the assessment, with one end representing "best imaginable health" and the other end representing "worst imaginable health."

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Zaragoza, Zaragoza, Aragon, Spain

IPD SHARING:
Plan to Share IPD: No